CLINICAL TRIAL: NCT04074824
Title: A Genome-Wide Association Study on Chinese Preterm Neonates and Identification of Functional Variants for Susceptibility to Necrotising Enterocolitis
Brief Title: A Genome-Wide Association Study for Neonatal Diseases
Status: Active, not recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Kathy Chan, Scientific Officer, Chinese University of Hong Kong
Other Study IDs: 2017.493
Record Dates: First submitted 2019-08-29; First posted 2019-08-30 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Neonatal Disease; Necrotizing Enterocolitis
MeSH Terms: conditions — Infant, Newborn, Diseases; Enterocolitis, Necrotizing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Buccal swabs and fecal samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Necrotizing enterocolitis: Neonates diagnosed with NEC based on the Modified Bell criteria for NEC including clinical, radiological and Laboratory findings.
- Non-NEC: Neonates diagnosed with other conditions including low birthweight, prematurity, infection, metabolic, cardiovascular, CNS, respiratory or gastrointestinal problems.

SUMMARY:
This is an observational study to identify genetic risks for neonatal diseases, necrotizing enterocolitis (NEC) using genome-wide association study (GWAS) and enterotype investigation. We hypothesize that specific genetic factors and microbiome could predispose preterm neonates for the development of NEC.

DETAILED DESCRIPTION:
NEC is the most frequently encountered surgical emergencies and a life-threatening disease that predominantly affects preterm neonates. The incidence is estimated to be 7-10% in ver low birth weight (VLBW) neonates (Lin and Stoll, 2006; Neu and Walker, 2011). However, a significant proportion of affected neonates (20-30%) develops severe progressive disease with intestinal necrosis and complications resulting in gut perforation and peritonitis which require urgent surgical intervention (surgical cases) (Sharma et al., 2006). The mortality rate of surgical cases is high (25-50%), and may increase to 100% in patients with pan-necrosis of the bowel. Those neonates who survived often suffer severe morbidity, including short bowel syndrome, parenteral nutrition-associated cholestasis, poor physical growth and neurodevelopmental impairment (Neu and Walker, 2011; Salhab et al., 2004). However, the etiology and pathophysiology of NEC remain incompletely understood. The current knowledge has directed towards multiple predisposing factors which include prematurity, immature gut mucosa and host defense immunity, formula milk feeding and altered microbial colonization in the gut resulting in excessive inflammatory response, leading to irreversible intestinal cell death and gut necrosis (Neu and Walker, 2011; Chan et al., 2013). To date, no genetic risk markers or biomarkers are available for reliable prediction of neonates who are at high risk of developing NEC. Besides host genetic factors, gut bacteria have been reported to predispose neonates to disease risk (Mai et. al., 2011; Neu and Pammi, 2018).

In this study, we shall conduct a GWAS on Chinese preterm neonates for identification of genetic risks for NEC and determine gut microbiome structure (enterotype) of NEC.

ELIGIBILITY:
Inclusion Criteria:

Chinese infants admitted in the neonatal unit (NNU)

Exclusion Criteria:

Refuse consent for study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Chinese infants
Sampling Method: Non-Probability Sample
Enrollment: 310 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
NEC | First year
  Neonatal Disease

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Chan, Ph. D., Principal Investigator — CUHK
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Background] Lin PW, Stoll BJ. Necrotising enterocolitis. Lancet. 2006 Oct 7;368(9543):1271-83. doi: 10.1016/S0140-6736(06)69525-1. PMID 17027734
- [Background] Neu J, Walker WA. Necrotizing enterocolitis. N Engl J Med. 2011 Jan 20;364(3):255-64. doi: 10.1056/NEJMra1005408. No abstract available. PMID 21247316
- [Background] Sharma R, Hudak ML, Tepas JJ 3rd, Wludyka PS, Marvin WJ, Bradshaw JA, Pieper P. Impact of gestational age on the clinical presentation and surgical outcome of necrotizing enterocolitis. J Perinatol. 2006 Jun;26(6):342-7. doi: 10.1038/sj.jp.7211510. PMID 16724075
- [Background] Salhab WA, Perlman JM, Silver L, Sue Broyles R. Necrotizing enterocolitis and neurodevelopmental outcome in extremely low birth weight infants <1000 g. J Perinatol. 2004 Sep;24(9):534-40. doi: 10.1038/sj.jp.7211165. PMID 15254558
- [Background] Chan KY, Leung KT, Tam YH, Lam HS, Cheung HM, Ma TP, Lee KH, To KF, Li K, Ng PC. Genome-wide expression profiles of necrotizing enterocolitis versus spontaneous intestinal perforation in human intestinal tissues: dysregulation of functional pathways. Ann Surg. 2014 Dec;260(6):1128-37. doi: 10.1097/SLA.0000000000000374. PMID 24368664
- [Background] Mai V, Young CM, Ukhanova M, Wang X, Sun Y, Casella G, Theriaque D, Li N, Sharma R, Hudak M, Neu J. Fecal microbiota in premature infants prior to necrotizing enterocolitis. PLoS One. 2011;6(6):e20647. doi: 10.1371/journal.pone.0020647. Epub 2011 Jun 6. PMID 21674011
- [Background] Neu J, Pammi M. Necrotizing enterocolitis: The intestinal microbiome, metabolome and inflammatory mediators. Semin Fetal Neonatal Med. 2018 Dec;23(6):400-405. doi: 10.1016/j.siny.2018.08.001. Epub 2018 Aug 17. PMID 30172660